CLINICAL TRIAL: NCT00841009
Title: Effect of Gastric Bypass-induced Weight Loss on Myocardial Structure, Function and Metabolism
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 05-0523
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Gastric Bypass
Keywords: gastric bypass; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 tubes of blood (1 tablespoon total) will be collected (with permission), tested and stored for a length of time
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity affects more than 43 million Americans and is associated with an increased incidence of heart failure, sudden death, and cardiovascular death. We have shown that increasing obesity is independently associated with potentially detrimental LV structural and functional, and metabolic changes. Thus in order to increase our understanding of the effect of obesity on the heart, we wish to study the effect of significant weight loss on these parameters.

DETAILED DESCRIPTION:
Thirty obese patients who weigh <350#, the weight limit of the PET table, who are to undergo gastric bypass will be enrolled in this study. Written, informed consent approved by the Institutional Review Board of Washington University School of Medicine will be obtained from each subject before his/her participation in this study. Subjects will be compensated for their time. Subjects will undergo Medical Screening (Visit 1) consisting of a comprehensive medical evaluation: a history (questionnaire), physical examination, EKG, blood chemistries, kidney function, complete blood count, lipid profiles and pregnancy tests for women of childbearing age. Subjects who weigh < 300# will have fat-free mass (body composition) determined by using a machine called DEXA. Measurement of Insulin Resistance (Visit 2): Subjects will undergo a hyperinsulinemic/euglycemic clamp and nonradiolabeled glucose infusion in order to define their level of insulin resistance and total body glucose turnover. This study will be performed in the GCRC.

Measurement of Myocardial Metabolism, Efficiency, Structure, and Function Measures and Total Body Fatty Acid Metabolism (Visit 3): Subjects will be admitted to the GCRC the evening before the PET imaging and at 6 pm will receive a standard meal. The next morning an 18-gauge intravenous catheter will be inserted into your arm vein. A catheter (small tube) will also be placed in the radial artery for the total body fat metabolism measurements & for blood pressure monitoring. If the subject wishes it, they may have a Foley placed for urination during the PET scan studies. Myocardial PET imaging. Studies will be performed during fasting conditions at 8 am and ending at 1:00 pm. Each subject will be positioned within the scanner, and a 2-min data collection will be acquired to verify proper positioning before a 5-min. scan will be performed for generation of attenuation correction factors. Heart blood flow, oxygen consumption, and measures of fat metabolism will be obtained using PET imaging after the sequential injections of radiolabeled tracers as reported previously by our group. Blood pressure and heart rate will be monitored continuously and recorded throughout the image acquisition. During the scans, 5 blood samples (0, 2, 10, 20,& 30 min) will be obtained for measurement of hormones, heart fuels (e.g. fats, lactate) and carbon dioxide levels.

Anonymous Genetic Tissue and Data Sampling: Draw and store 1 tablespoon of subject's blood, for a period of up to 10 years, to be used in future studies for screening for differences in genes related to heart membrane proteins or heart energy metabolism (including but not limited to genes known as KV1.5, KV2.1, PPAR, FATP, ACS, PGC-1). Echocardiography: Immediately following the PET imaging for oxygen consumption determination, subjects will undergo a complete 2D-, 3D-, and Doppler echocardiographic examination. Optison or Definity, depending on availability, clinically used intravenous contrast agents may be administered to aid with the acquisition of the ultrasound images. Total body fatty acid metabolism measurements: Simultaneous with the PET imaging, the subjects will undergo an infusion of a tracer amount of nonradioactive fat for measurement of total body fat metabolism. Blood samples will be drawn at predetermined times for this measurement.

3 Months s/p Gastric Bypass Surgery (Visit 4). Blood sampling

1 Year s/p Gastric bypass Measurement of Body Composition, Blood Chemistries, Lipid Levels, and Insulin Resistance (Visits 5 and 6). After the subjects have undergone gastric bypass for clinical reasons and are weight stable for 2 weeks (after approximately 1 year post-gastric bypass).

ELIGIBILITY:
Inclusion Criteria:

* Subjects that will undergo gastric bypass surgery will be included in the study.

Exclusion Criteria:

* Subjects who have a history of insulin-requiring diabetes, ≥Class II hypertension, cardiac disease, major systemic disease, of smoking cigarettes with in the last 12 months, who are pregnant or taking vasoactive or lipid-lowering medications will be excluded because these conditions may affect our cardiac endpoints. Subjects unable to give informed consent will be excluded. Subjects > 350# (the weight limit of the PET table) will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who are to undergo gastric bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2005-07; Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
measure the effect of marked weight loss induced by gastric bypass surgery on myocardial metabolism, efficiency, structure, and function in morbidly obese men and women | measure at year 5

SECONDARY OUTCOMES:
evaluate the relationship between changes in myocardial lipid metabolism with changes in whole-body lipid metabolism caused by weight loss | measure at year 5

CONTACTS AND LOCATIONS:
Overall Officials: Linda Peterson, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Bergman RN, Ider YZ, Bowden CR, Cobelli C. Quantitative estimation of insulin sensitivity. Am J Physiol. 1979 Jun;236(6):E667-77. doi: 10.1152/ajpendo.1979.236.6.E667. PMID 443421
- [Background] Pacini G, Bergman RN. MINMOD: a computer program to calculate insulin sensitivity and pancreatic responsivity from the frequently sampled intravenous glucose tolerance test. Comput Methods Programs Biomed. 1986 Oct;23(2):113-22. doi: 10.1016/0169-2607(86)90106-9. PMID 3640682
- [Background] Young ME, Razeghi P, Cedars AM, Guthrie PH, Taegtmeyer H. Intrinsic diurnal variations in cardiac metabolism and contractile function. Circ Res. 2001 Dec 7;89(12):1199-208. doi: 10.1161/hh2401.100741. PMID 11739286
- [Background] Kates AM, Herrero P, Dence C, Soto P, Srinivasan M, Delano DG, Ehsani A, Gropler RJ. Impact of aging on substrate metabolism by the human heart. J Am Coll Cardiol. 2003 Jan 15;41(2):293-9. doi: 10.1016/s0735-1097(02)02714-6. PMID 12535825
- [Background] Bergmann SR, Herrero P, Markham J, Weinheimer CJ, Walsh MN. Noninvasive quantitation of myocardial blood flow in human subjects with oxygen-15-labeled water and positron emission tomography. J Am Coll Cardiol. 1989 Sep;14(3):639-52. doi: 10.1016/0735-1097(89)90105-8. PMID 2788669
- [Background] Herrero P, Markham J, Bergmann SR. Quantitation of myocardial blood flow with H2 15O and positron emission tomography: assessment and error analysis of a mathematical approach. J Comput Assist Tomogr. 1989 Sep-Oct;13(5):862-73. doi: 10.1097/00004728-198909000-00021. PMID 2789240
- [Background] Herrero P, Hartman JJ, Senneff MJ, Bergmann SR. Effects of time discrepancies between input and myocardial time-activity curves on estimates of regional myocardial perfusion with PET. J Nucl Med. 1994 Apr;35(4):558-66. PMID 8151375